CLINICAL TRIAL: NCT06041308
Title: Long-term Outcomes of Bioprothetic Valve Versus Mechanical Valve
Brief Title: Bioprothetic Valve Versus Mechanical Valve of Bioprothetic Valve Versus Mechanical Valve
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012072RIND
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-03

CONDITIONS: Valve Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bioprothetic valve: Groups undergoing cardiac valve surgery with bioprothetic valve.
  Interventions: Other: valve
- Mechanical valve: Groups undergoing cardiac valve surgery with mechanical valves.
  Interventions: Other: valve

INTERVENTIONS:
Other: valve — bioprothetic valve versus mechanical valve

SUMMARY:
In this study, the investigators aim to use data identified through the hospital's integrated medical database and National Health Insurance database to explore the long-term performance and benefits of biological and mechanical valves. This research aims to provide more recommendations and references for valve replacement in different patient populations.

DETAILED DESCRIPTION:
Long-term follow-up of valve surgery is essential in all cardiac surgeries and is the most commonly discussed indicator. The choice of valves has evolved over the past 30 years, offering two options: biological valves and mechanical valves. Biological valves have seen advancements in the last 15 years, including new processes and improved valve preservation methods. The question of whether these new process valves offer better long-term effectiveness has become a hot research topic in recent years.

Mechanical valves have a longer lifespan, but the need for long-term anticoagulant use to prevent mechanical valve thrombosis has raised concerns about anticoagulant side effects, abnormal clotting function, and bleeding. Biological valves, on the other hand, do not require long-term anticoagulation and only necessitate 2-3 months of anticoagulant treatment. However, the risk of biological valve degeneration results in an average lifespan of 10 to 20 years, which cannot match the durability of mechanical valves. This is the drawback of using biological valves.

Therefore, the investigators hope to utilize the hospital's integrated medical database and the long-term National Health Insurance database for tracking. The investigators aim to observe valve performance in different patient groups, such as young people, the elderly, patients on dialysis, those with rheumatic autoimmune diseases, and those taking specific medications, among others.

ELIGIBILITY:
Inclusion Criteria:This is a retrospective study, and we plan to utilize data from the hospital's integrated medical database and the National Health Insurance database from January 2007 to December 2019. We will identify all patients within the data who were diagnosed with valve diseases and underwent valve replacement surgery.

-

Exclusion Criteria:Individuals under 20 years of age.

-

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 30,000 individuals (including this institution and other domestic units).
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 1998-2019
  included estimated survival using a Cox regression model. Survival data were obtained for all NHIRD databases. Operative mortality was defined as death during the index hospitalization or within 30 days of the operation. Long-term survival data included death from all causes.
  survival outcome was measured months after the index operation.

SECONDARY OUTCOMES:
composite outcome and individual component of major adverse prosthesis-related events, including death, major bleeding, ischemic stroke, endocarditis, and aortic valve reoperation | 1998-2019
  each of which were defined as an emergency room visit or hospital admission with related diagnosis codes as the primary diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Hsin Chi, Study Chair — attending physician
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Takei Y, Chou NK, Wei LY, Fu HY, Yu HY, Chi NH. Robotic transmitral approach in hypertrophic cardiomyopathy. Int J Surg. 2024 Nov 1;110(11):7391-7394. doi: 10.1097/JS9.0000000000001934. No abstract available. PMID 38995189